CLINICAL TRIAL: NCT07095010
Title: Evaluation of the Role of Lifestyle Habits in the Presence of Metabolic Dysfunction-associated Steatotic Liver Disease in a Sample of Greek Children and Adolescents
Brief Title: Lifestyle Habits and Metabolic Dysfunction-Associated Steatotic Liver Disease in Youth
Acronym: LIFE4MASLD
Status: Completed | Type: Observational
Sponsor: Harokopio University (Other)
Collaborators: Children 's Hospital, Agia Sophia (Unknown)
Responsible Party: Principal Investigator, Meropi Kontogianni, Professor of Clinical Nutrition, Harokopio University
Other Study IDs: 5296
Record Dates: First submitted 2025-06-06; First posted 2025-07-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The following samples will be retained and stored at -80°C: 2 ml of serum, 2 ml of plasma, and 2 ml of urine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is the most common cause of chronic liver disease in children and adolescents. Lifestyle factors are modifiable risk factors that may play a key role in both the prevention and management of the disease. However, existing data on the association between lifestyle and MASLD in pediatric populations are limited and often focus on isolated aspects such as diet or physical activity, with little attention given to other parameters like sleep habits. The aim of the present study is to comprehensively investigate the association between lifestyle factors, including dietary habits, physical activity, sedentary activities, and sleep habits, and the presence of MASLD in a sample of 224 children and adolescents with overweight or obesity. The study will include newly diagnosed MASLD patients compared to matched controls without the disease. A wide range of assessments will be conducted, including anthropometric measurements, body composition analysis, liver elastography, biochemical testing, and standardized lifestyle questionnaires. This study seeks to fill important research gaps and explore potential associations between lifestyle habits and pathophysiological markers involved in the onset and progression of MASLD.

DETAILED DESCRIPTION:
The study sample will consist of 224 children and adolescents aged 10-18 years with overweight or obesity, including individuals newly diagnosed with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) and matched controls without the disease.

The diagnosis of MASLD will be based on the criteria established by the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN): elevated alanine aminotransferase (ALT) levels >45 IU/L and/or evidence of hepatic steatosis on ultrasound, in the absence of other causes of liver steatosis or liver injury. Where available, liver biopsy results will be included in the participants' medical records.

Participants in the control group will be matched to the MASLD group based on age, sex, body mass index (BMI), and pubertal stage. Eligible controls must present with normal liver biochemistry, no ultrasound evidence of hepatic steatosis, normal glucose metabolism, and stable body weight and lifestyle behaviors during the past year.More specifically, the study will include:

1. Medical and family history: Detailed documentation of personal and family medical history, current medications, and birth-related data (e.g., gestational age, birth weight, breastfeeding history).
2. Demographic and socioeconomic data: Collected from both parents and participants, including education level, employment status, ethnicity, and household composition.
3. Anthropometric measurements and body composition: Body weight, height, BMI, waist and hip circumference will be recorded. Body composition will be assessed using bioelectrical impedance analysis (Tanita MC 780 MA), with standardized conditions (e.g., fasting state, no intense physical activity, no caffeine intake).
4. Blood pressure: Measured in a seated position with an electronic sphygmomanometer on the right arm. Three measurements will be taken, and the mean value will be recorded.
5. Liver imaging: All participants will undergo abdominal ultrasound for assessment of hepatic steatosis, and those with MASLD will undergo liver elastography (Shear Wave Elastography) within 3 months of enrollment to evaluate liver fibrosis.
6. Laboratory testing: After 8-12 hours of fasting, blood samples will be collected to determine standard biochemical profile, including liver enzymes (ALT, AST, GGT), bilirubin, lipids (total cholesterol, HDL, LDL, triglycerides), glucose, insulin, kidney function, electrolytes, and total protein, hematologic markers (complete blood count and erythrocyte sedimentation rate), inflammation and oxidative stress biomarkers, and oxidative stress markers. Serum, plasma, and urine samples will be stored at -80°C for future analyses. DNA will also be extracted for potential genotyping.
7. Fatty Liver Index (FLI): FLI will be calculated using waist circumference, BMI, triglyceride levels, and GGT to assess the risk of hepatic steatosis.
8. Dietary assessment: Each participant will complete four 24-hour dietary recalls (three weekdays and one weekend day). Nutrition data will be analyzed for energy, macro- and micronutrient intake using Nutritionist Pro (v2.2), with additional assessment of food groups and dietary patterns. Adherence to the Mediterranean Diet will be assessed using the KIDMED index.
9. Physical activity assessment: Performed using the Self-Administered Physical Activity Checklist (SAPAC), validated for the Greek pediatric population. It will be completed four times, in conjunction with the dietary recalls.
10. Sleep habits assessment: Evaluated with the Pediatric Daytime Sleepiness Scale (PDSS), along with additional questions about sleep duration, naps, and rest habits on weekdays and weekends.

ELIGIBILITY:
Inclusion Criteria:

* Age: Children and adolescents aged 10 to 18 years, of Caucasian ethnicity, regardless of sex or nationality.
* Overweight or Obesity: Children/adolescents with overweight or obesity according to World Health Organization (WHO) criteria for ages 5-19.
* Newly Diagnosed Metabolic Dysfunction-Associated Steatotic Liver Disease: Diagnosis will be established in participants who meet all of the following criteria:

  * Elevated ALT levels (>45 IU/L), according to the European Society for Paediatric Gastroenterology, Hepatology and Nutrition, and/or evidence of hepatic steatosis on liver ultrasound.
  * Exclusion of other causes of liver damage or steatosis, including negative for HBsAg, anti-HIV, and anti-HCV antibodies, no autoimmune hepatitis, no viral infections, systemic or metabolic diseases, no celiac disease, chronic kidney disease, normal ceruloplasmin levels (to rule out Wilson's disease), no hepatotoxic medications.

Exclusion Criteria:

* Type 1 diabetes mellitus
* Alcohol consumption
* Malnutrition or parenteral nutrition
* Thyroid function
* Recent changes in diet and physical activity habits aimed at weight loss and/or improvement of health parameters in newly diagnosed children and adolescents

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 224 children and adolescents with overweight/ obesity and/or Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Differences in dietary intake between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  The dietary intake of the participants will be assessed by four 24-hour recall method and analyzed using the Nutritionist Pro software program.
Difference in adherence to the Mediterranean diet between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  The adherence to the Mediterranean diet will be evaluated using the KIDMED questionnaire. The index of adherence to the Mediterranean diet was calculated as the sum of each answer and ranged from 0 to 12. The sums of the values of the KIDMED score will be classified into three levels: (1) >8, optimal Mediterranean diet; (2) 4-7, improvement needed to adjust intake to Mediterranean patterns; (3) ≤3, very low diet quality.
Differences in physical activity between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  Physical activity will be assessed using the Self-Administered Physical Activity Checklist, a questionnaire validated in the Greek population. This checklist records the type, frequency, and duration of physical activities performed in the previous day. Each participant (or their caregiver) will complete the checklist four times, with the assistance of a registered dietitian, immediately following the 24-hour dietary recall interviews.
  From the collected data, the average daily time spent in physical activity (in minutes per day) will be calculated. The checklist yields a quantitative score ranging from 0 to an unlimited maximum, depending on the number and duration of activities reported. Higher scores indicate greater levels of physical activity, reflecting more time spent in moderate-to-vigorous physical activity during the assessed day.
Differences in sedentary activities between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  Sedentary activities will be assessed with the Self-Administered Physical Activity Checklist (SAPAC), a questionnaire validated for the Greek population. Each participant (or caregiver) will complete the checklist four times with support from a registered dietitian immediately after each 24-hour dietary recall.
  For every administration, the SAPAC records the duration of common sedentary behaviours (e.g., television viewing, videogaming, seated reading). The summed sedentary-time score is expressed in hours per day and has a possible range of 0 h (no sedentary time) to 24 h (continuous sedentary behaviour). Higher scores indicate a worse outcome, namely, more time spent in sedentary activities. The mean of the four administrations will be used as each participant's average daily sedentary time.
Differences in sleep hours between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  Total night sleep hours will be recorded.
Differences in daytime sleepiness between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. | Baseline
  The daytime sleepiness will be evaluated using the Pediatric Daytime Sleepiness Scale (score range 0-32). Higher scores indicated greater levels of sleepiness.

SECONDARY OUTCOMES:
hs-CRP | Baseline
  Differences in hs-CRP between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. hs-CRP (mg/L) will be measured via nephelometry (BN II nephelometer, Siemens).
Adiponectin | Baseline
  Differences in adiponectin between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. Adiponectin (μg/mL) will be quantified using immunoenzymatic ELISA kits (Human Adiponectin ELISA Kit).
Fibroblast Growth Factor 21 | Baseline
  Differences in Fibroblast Growth Factor 21 (FGF-21) between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. FGF-21 (pg/mL) will be quantified using immunoenzymatic ELISA kits (Human Total FGF-21 Quantikine, R&D Systems).
Oxidative stress | Baseline
  Differences in oxidative stress between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. Oxidative stress will be assessed by measuring serum TBARS (μM) using a modified colorimetric assay.
Insulin resistance | Baseline
  Differences in insulin resistance between children and adolescents with overweight/obesity and MASLD and their matched controls without MASLD. Insulin resistance will be assessed using the HOMA-IR index, calculated as [fasting glucose (mmol/L) × insulin (μU/mL)] / 22.5, as proposed by Matthews et al.

CONTACTS AND LOCATIONS:
Overall Officials: Meropi D Kontogianni, Principal Investigator — Harokopio University Athens, Kallithea, Greece
Locations (1):
- Harokopio University, Athens, Kallithea, Greece